CLINICAL TRIAL: NCT03796377
Title: Effects of Hypericum Perforatum (St. John's Wort) on the Pharmacokinetics and Pharmacodynamics of Rivaroxaban in Humans
Brief Title: Rivaroxaban Hypericum Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: Studien-Nr. 3459
Record Dates: First submitted 2019-01-04; First posted 2019-01-08 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Drug Interaction Study
MeSH Terms: interventions — Hypericum extract LI 160; ATP Binding Cassette Transporter, Subfamily B, Member 1; Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rivaroxaban (Other): Single oral dose of 20 mg rivaroxaban
  Interventions: Drug: Rivaroxaban
- Rivaroxaban after CYP- and P-gp induction (Other): Single oral dose of 20 mg rivaroxaban after pretreatment with St. John's wort extract (Jarsin®) twice daily 450 mg po for 2 weeks.
  Interventions: Drug: St Johns Wort Extract; Drug: Rivaroxaban

INTERVENTIONS:
Drug: St Johns Wort Extract — 20 mg rivaroxaban after supplementation with St. John's wort extract (Jarsin®) twice daily 450 mg po for 2 weeks.
  Other Names: Inducer of CYP3A4 and P-gp
  Arms: Rivaroxaban after CYP- and P-gp induction
Drug: Rivaroxaban — 20 mg rivaroxaban.

SUMMARY:
Single-center, open-label, sequential treatment study to investigate the influence of the combined P-glycoprotein and CYP3A4 inducer hypericum perforatum on the pharmacokinetics and pharmacodynamics of rivaroxaban in healthy volunteers.

DETAILED DESCRIPTION:
Each session (one with and one without preceding CYP induction) will start with phenotyping using 25 mg fexofenadine orally for P-gp phenotyping and 2 mg midazolam orally for cytochrome P450 (CYP) 3A4 phenotyping. After a washout period of 5 days, subjects will receive a single oral dose of 20 mg rivaroxaban, a dose currently approved for human use in clinical routine. The same procedure will be repeated after pretreatment with St. John's wort extract (Jarsin®) twice daily 450 mg po (dose usually used in clinical routine) for 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, age between 18 and 45 years (inclusive) at screening
* BMI between 18 and 28 kg/m2 (inclusive) at screening
* No clinically significant findings on the physical examination at screening
* Hematology and clinical chemistry results not deviating from the normal range to a clinically relevant extent at screening
* Ability to communicate well with the investigator and to understand and comply with the requirements of the study
* Women of child-bearing age: willingness of using a double barrier contraception method during the study, i.e. a hormonal method (oral contraceptive, intrauterine device) in combination with a mechanical barrier (e.g. condom, diaphragm)
* Signed informed consent

Exclusion Criteria:

* Known allergic reaction to any excipient of the drug formulations
* Known photosensitivity
* Smoking
* History or clinical evidence of alcoholism or drug abuse within the 3-year period prior to screening
* Loss of ≥ 250 ml of blood within 3 months prior to screening, including blood donation
* Treatment with an investigational drug within 30 days prior to screening
* Previous treatment with any prescribed or over-the-counter medications (including herbal medicines such as St. John's wort) within 2 weeks prior to screening
* Pregnant (positive results from urine drug screen at screening) or lactating women
* History or clinical evidence of any disease (e.g. gastrointestinal tract disease) and/or existence of any surgical or medical condition, which might interfere with the absorption, distribution, metabolism or excretion of the study drugs, or which might increase the risk for toxicity
* Legal incapacity or limited legal capacity at screening
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2019-04-09 (Actual); Study Completion 2019-04-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic outcome measures: area under the curve (AUC). | AUC will be calculated from the concentration-time plot (time points included: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, and 48 hours (post-dose) during both sessions)
  Effect of pretreatment with hypericum perforatum on geometric mean AUC.
Pharmacokinetic outcome measures: maximal concentration of rivaroxaban. | Will be obtained from the individual plasma concentration data (time points included: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, and 48 hours (post-dose) during both sessions)
  Effect of pretreatment with hypericum perforatum on maximal concentration of rivaroxaban.
Pharmacodynamic outcome measures: Factor Xa activity | Time points used for analysis: pre-dose, 0.5, 1, 2, 4, 8, 12, 24, 36, and 48 hours (post-dose) during both sessions
  Displayed as maximal effect (Emax) and parametrized by calculating the area under the time-effect curves (AUEC)).

SECONDARY OUTCOMES:
Pharmacokinetic parameters: Time to reach maximal concentration | Time points used for analysis: 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, and 48 hours (post-dose) during both sessions
  Time to reach maximal concentration of rivaroxaban
Pharmacokinetic parameters: Plasma elimination half-life | Time points used for analysis: 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, and 48 hours (post-dose) during both sessions
  Plasma elimination half-life of rivaroxaban
Phenotyping metrics: AUC fexofenadine | Time points used for analysis: Before dosing and 0.5, 2, 3, 6 h after administration
  Estimated AUC of fexofenadine
Phenotyping metrics: AUC ratios midazolam | Time points used for analysis: Before dosing and 0.5, 2, 3, 6 h after administration
  AUC ratios of midazolam and 1'-hydroxymidazolam
Phenotyping metrics: Single point metabolic ratios midazolam | Time points used for analysis: Before dosing and 0.5, 2, 3, 6 h after administration
  Single point metabolic ratios of midazolam and 1'-hydroxymidazolam

CONTACTS AND LOCATIONS:
Overall Officials: Inselpital, Study Director — Sponsor: Inselspital, Bern University Hospital
Locations (1):
- Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Scholz I, Liakoni E, Hammann F, Grafinger KE, Duthaler U, Nagler M, Krahenbuhl S, Haschke M. Effects of Hypericum perforatum (St John's wort) on the pharmacokinetics and pharmacodynamics of rivaroxaban in humans. Br J Clin Pharmacol. 2021 Mar;87(3):1466-1474. doi: 10.1111/bcp.14553. Epub 2020 Oct 25. PMID 32959922